CLINICAL TRIAL: NCT07203313
Title: Development, Feasibility, and Acceptability of Aim to Play, a User-Friendly Digital Application for Teacher Skills Training and Physical Education Activities for 3-5 Grade Elementary Students
Brief Title: Evaluation of Aim to Play, a User-Friendly Digital Application for Teacher Skills Training and Physical Education Activities for 3-5 Grade Students
Acronym: AimToPlay3-5
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saavsus, Inc. (Other)
Collaborators: Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R44DP006743 (NIH); R44DP006743 (NIH)
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Teacher Self-efficacy for Teaching PE; Teacher PE Instruction; Student PE Enjoyment; Student Physical Activity; Student PE Satisfaction
Keywords: physical activity; physical education; elementary school; children
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pocket PE 3-5 (Experimental)
  Interventions: Behavioral: Digital PE teaching app
- Business as usual (No Intervention): Control group

INTERVENTIONS:
Behavioral: Digital PE teaching app — Pocket PE 3-5 is a digital app designed for 3rd - 5th grade teachers and students. It works across common platforms and devices, online and offline, and provides simple, easy to use, standards-based PE lesson activities tailored by time, instructional setting (classroom, gym, outside), grade, student skill level, and equipment resources. The app is low-cost and includes brief teacher and student skill demonstration videos for each activity, along with printable activity cards, music, and audio cues to signal transitions to assist teachers in class management with students in real time during PE. The program also includes embedded data tracking of PE minutes and completed instructional standards to assist with school and/or state mandated reporting.
  Other Names: Pocket PE 3-5; Aim to Play 3-5
  Arms: Pocket PE 3-5

SUMMARY:
The goal of this clinical trial is to evaluate the newly developed Pocket PE 3-5 app, designed for use by teachers of 3rd-, 4th-, and 5th-grade students. Researchers will compare teachers and students in classrooms using the Pocket PE app with those in classrooms not using the app.

The main question it aims to answer is:

• Does the use of the Pocket PE 3-5 app improve classroom teacher PE self-efficacy and high-quality PE teaching behaviors, and promote students' moderate-to-vigorous physical activity participation in PE, as well as PE enjoyment and self-efficacy, compared to teachers who do not use Pocket PE 3-5?

Participants will:

* Randomly use Pocket PE 3-5 (12 intervention schools) for at least one PE class weekly, or not (12 control schools), for 12 consecutive weeks during the 2025/26 school year.
* Teachers will complete short surveys at 0 weeks (pre), 6 weeks (mid), and 13 weeks (post). Teachers in the intervention condition will complete a longer survey at 13 weeks (post-intervention) to provide feedback on the Pocket PE app. A random sub-sample of teachers in the intervention condition will be asked to participate in an exit interview to give additional input on Pocket PE 3-5 after the intervention has been completed.
* Students will complete brief surveys after PE classes at pre, mid, and post, and will wear wrist heart rate monitors during observed PE classes at these timepoints to measure their physical activity during PE.

We will also evaluate the level of implementation of Pocket PE 3-5 among teachers via class observations and objective data collected by the app.

DETAILED DESCRIPTION:
Childhood physical inactivity is associated with a myriad of preventable health inequities among children, including greater prevalence and more severe childhood obesity, poorer cardiovascular and bone health, and lower levels of cognitive functioning, mental health, and self-esteem. While 43 states currently have laws mandating elementary school physical education (PE) to promote student public health objectives, most students do not achieve adequate PE participation because teachers (both PE certified and regular classroom teachers or paraprofessionals who teach PE) have limited or no access to easy-to-use and low-cost programmatic resources that address salient barriers for conducting effective, evidence-based, and standards-based PE.

The Pocket PE 3-5™ digital app (initially conceptualized as Aim to Play 3-5TM) is designed for 3rd - 5th grade teachers and students and works across common platforms and devices, online and offline, and provides simple, easy to use, standards-based PE lesson activities tailored by time, instructional setting (classroom, gym, outside), grade, student skill level, and equipment resources. The app is low-cost and includes brief teacher skill demonstration videos for each activity, along with printable activity cards, music, and audio cues to signal transitions to assist teachers and students with class management in 'real time' during PE. The program also includes embedded data tracking of PE minutes and completed instructional standards to assist with district and/or state-mandated reporting. Pocket PE 3-5 offers a technology-driven solution to promote the adoption of Comprehensive School Physical Activity Programs (CSPAPs) by providing a scalable, evidence-based resource to schools to promote high-quality PE participation among students.

To evaluate Pocket PE 3-5, we will conduct a cluster-randomized trial in 24 elementary schools, with one identified 3rd-, 4th-, and 5th-grade classroom teacher and their students in each school. Participating schools will be in California and Oregon and will be randomly assigned to receive Pocket PE 3-5 (n = 12 intervention schools) or not (n = 12 control schools) over a 12-week period. We anticipate that 72 teachers and approximately 1,800 students will participate. Assessments at pre, mid, and post program will primarily occur at the teacher level on PE class instruction, fidelity of implementation, and PE teaching self-efficacy. Teachers using Pocket PE (assigned to the intervention condition) will also provide feedback on the app, including usability, acceptability, and satisfaction. We will explore secondary student outcomes focused on objectively measured minutes of moderate-to-vigorous physical activity achieved during PE and PE enjoyment, as well as program satisfaction and enjoyment.

Hypothesis: Intervention teachers will improve their PE teaching self-efficacy and teaching practices, and students will participate in more moderate-to-vigorous physical activity during PE and have greater PE enjoyment and satisfaction, relative to the control group.

ELIGIBILITY:
Inclusion Criteria for teachers:

* A 3rd, 4th, or 5th grade teacher at a participating school responsible for teaching PE at least one time a week;
* Able to read and understand English;
* Willing to use Pocket PE to facilitate their PE class instruction for 12 weeks;
* Be able to understand the study and consent to participate

Inclusion Criteria for students:

* A 3rd, 4th, or 5th grader enrolled in a participating class in a participating school;
* Able to read and understand English;
* Able to understand the study and assent to participation;

Exclusion Criteria:

* None

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1872 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Teaching Physical Activity (PE) Self Efficacy | Pre (0 weeks), mid (6 weeks after pre), and post (13 weeks after pre)
  This is a 20-item survey assessing the self-efficacy for PE instruction scale, adapted from Humphries, Daigle, & Martin (2012). Each item is on a 10-point scale (1 = disagree/cannot do, 5 = neutral/moderate certainty, 10 = agree/highly certain can do). Items are summed for a score that can range from 20 to 200, with a higher score indicating higher levels of teacher physical activity self-efficacy.
System for Observing Fitness Instruction Time (SOFIT) | Pre (0 weeks), mid (6 weeks after pre), and post (13 weeks after pre)
  The SOFIT assesses physical education classes by obtaining simultaneous, objective observational data on student activity levels, the context in which they occur, and how teachers interact to promote physical activity and fitness during physical education. Student activity levels include the percent of time a student is in moderate-to-vigorous physical activity (% MVPA = intervals with codes 4 or 5) ÷ (total intervals) × 100) and percent of time the student is in vigorous activity (% VA = %VPA = (intervals with code 5) ÷ (total intervals) × 100). Interval 4 = walking/moderate, and interval 5 = vigorous. The context in which the activity can occur is summarized at a percentage of time in: M (general content: management/transition/break), K (knowledge), and the motor-content categories F (fitness), S (skill practice), G (game play), O (other/free play).

SECONDARY OUTCOMES:
Student physical activity | Pre (0 weeks), mid (6 weeks after pre), and post (13 weeks after pre)
  Students will wear heart rate wrist monitors during an observed PE class to assess activity levels. The total number of minutes of moderate-to-vigorous physical activity will be computed from the heart rates.
Student PE Enjoyment | Pre (0 weeks), mid (6 weeks after pre), and post (13 weeks after pre)
  This is a single-item scale created by the study asking students, "How did you like PE today?". The response option is on a 5-point scale, where 1 = 'not at all' and 5 = 'a lot'. A higher score indicates greater enjoyment of PE.
Student PE Self-Efficacy | Pre (0 weeks), mid (6 weeks after pre), and post (13 weeks after pre)
  This is a 4-item self-efficacy scale developed by Morano, Bortoli, Ruiz, Vitali, & Robazza (2019). Students are asked, "When I do PE at school:" and there are four response options, each with a different set of responses. For example, for one item 1 = "I run very slowly" and 5 = "I run very fast". A mean score is computed and can range from 1 to 4. A higher score indicates higher levels of student PE self-efficacy.
Student PE Enjoymnet | Pre (0 weeks), mid (6 weeks after pre), and post (13 weeks after pre)
  This is a 4-item PE enjoyment scale developed by Morano, Bortoli, Ruiz, Vitali, & Robazza (2019). There are 4 items, and each item has a 5-point response option (1 = not at all, 5 = very much). A mean score is computed and can range from 1 to 5. A higher score indicates higher levels of PE enjoyment.

OTHER OUTCOMES:
Usefulness of the Pocket PE app features | Post (13-weeks after Pre)
  This is a 9-item scale created by the study team for this study. The items assessed teacher ratings of how useful they thought the Pocket PE App features were (e.g., inputting lesson parameters, viewing activity illustrations). The items are evaluated with a 5-point response option (1 = not at all useful, 5 = extremely useful). A mean score is computed and can range from 1 to 5, and a higher score indicates higher levels of perceived usefulness of the app.
Pocket PE App as a Resource for Teaching PE | Post (13-weeks after Pre)
  This is an 8-item scale created by the study team for this study. The items assess teacher ratings of the Pocket PE App as a resource for teaching RE (e.g., help start the PE session quickly). The items are evaluated with a 5-point response option (1 = strongly disagree, 5 = strongly agree). A mean score is computed and can range from 1 to 5, and a higher score indicates higher levels of satisfaction with the app as a resource for teaching PE.
Pocket PE App System Usability Scale | Post (13-weeks after Pre)
  This is a 10-item adaptation of the System Usability Scale (SUS; Brooke, 1996) which measures how well teachers rate the usability of the Pocket PE app (e.g., I thought the Pocket PE app was easy to use). Response options are on a 5-point scale, ranging from 1 (strongly disagree) to 5 (strongly agree). For odd-numbered items, the value of 1 is subtracted from the score, and for even-numbered items, the response is subtracted from 5. Items are then summed and multiplied by 2.5. Total scores can range from 0 to 100, with higher scores indicating higher levels of usability.
Pocket PE App Acceptability Rating | Post (13-weeks after Pre)
  This is a 7-item scale adapted from the Acceptability factor from the Behavior Intervention Rating Scale (Elliott & Treuting, 1991). Response options are on a 5-point scale from 1 (strongly disagree) to 5 (strongly agree). A mean score is computed across all items and can range from 1 to 5. A higher score indicates higher levels of app acceptability.
Helpfulness of the Pocket PE App | Post (13-weeks after Pre)
  This is a 7-item scale created by the study team for this study. The items assess teacher ratings of how helpful they thought the Pocket PE App was (e.g., Planning PE classes, managing student activity). The items are evaluated with a 5-point response option (1 = not at all helpful, 5 = extremely helpful). A mean score is computed and can range from 1 to 5, and a higher score indicates higher levels of perceived helpfulness of the app.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Saavsus, Inc., Eugene, Oregon
  - Oregon Research Institute, Springfield, Oregon

IPD SHARING:
Plan to Share IPD: Yes